CLINICAL TRIAL: NCT02690311
Title: A Study on the Changes of the Biological Rhythm by Display Image Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2013-08-072
Record Dates: First submitted 2016-01-28; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2013-08

CONDITIONS: Circadian Rhythm Phase Shift

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LED with bluelight (Sham Comparator): Two types of smartphone were used. One type had a conventional LED display with the full range of blue light. The LED in the other type newly developed by Samsung Display was suppressed for the blue light portion of the spectrum (wavelength 450 ~ 470 nm). The smartphones were indistinguishable from each other with the naked eye, because other wavelengths mimicked blue light in the suppressed LED.
  Interventions: Device: smartphone display
- LED without bluelight (Experimental): Two types of smartphone were used. One type had a conventional LED display with the full range of blue light. The LED in the other type newly developed by Samsung Display was suppressed for the blue light portion of the spectrum (wavelength 450 ~ 470 nm). The smartphones were indistinguishable from each other with the naked eye, because other wavelengths mimicked blue light in the suppressed LED.
  Interventions: Device: smartphone display

INTERVENTIONS:
Device: smartphone display

SUMMARY:
Effects of Smartphone Use at Night with Light Emitting Diode Display With and Without Blue Light in Healthy Adults: A Randomized, Double-blind, Cross-over, Placebo-controlled Comparison

ELIGIBILITY:
Inclusion Criteria:

(1) Healthy males 20-40 years of age who understood the study procedure and agreed to participate after being fully informed about the study were included.

Exclusion Criteria:

1. psychiatric diseases according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria;15
2. cognitive or neurological disorders;
3. alcohol or substance abuse;
4. unstable or serious medical illness;
5. current use of psychoactive mediations including antidepressants, anxiolytics, neuroleptics, anticonvulsants, hypnotics, or stimulant medications;
6. primary sleep disorder;
7. habitual sleep onset earlier than 21:00 or later than 24:00;
8. shift worker;
9. travel across more than two time zones within 90 days of the study; and
10. ophthalmologic disease during the study period.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes of serum melatonin | serum melatonin levels were measured every 60 min from 7:00 PM on day 1 to 8:00 AM on day 2, from 7:00 PM on day 2 to 8:00 AM on day 3, and from 7:00 PM to 11:00 PM on day 3 for 3 days.
Changes of serum cortisol | cortisol levels were measured every 120 min from 7:00 PM on day 1 to 8:00 AM on day 2, from 7:00 PM on day 2 to 8:00 AM on day 3, and from 7:00 PM to 11:00 PM on day 3 for 3 days.
Changes of body temperature | body temperature was measured every 120 min from 7:00 PM on day 1 to 8:00 AM on day 2, from 7:00 PM on day 2 to 8:00 AM on day 3, and from 7:00 PM to 11:00 PM on day 3 for 3days.

SECONDARY OUTCOMES:
profile of mood states(POMS) | day 1,3
  Mood was measured using the POMS,17 a well-validated self-report measure of mood states.
Epworth Sleepiness Scale(ESS) | day 1,3
  ESS18 is comprised of eight questions that query the subject's likelihood of dozing off or falling asleep in a particular situation that is commonly met in daily life.
Fatigue severity scale(FSS) | day 1,3
  The FSS20 is composed of 9 statements (items) that describe fatigue symptoms. Respondents select the most relevant level of agreement over the last week on a 7-point scale (1 strongly disagree; 7 strongly agree).
continuous performance test(CPT) | day1,3
  Integrated visual-auditory CPTs were performed at days 1 and 3 by a psychologist who was an expert on cognitive tests